CLINICAL TRIAL: NCT01366456
Title: Clinical Trials for Comparison Between Shingigu and Charcoal Moxa on CV-12
Brief Title: Clinical Trials for Comparison of Two Kinds of Moxibustion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semyung University (Other)
Collaborators: Kyunghee University (Other)
Responsible Party: Hoyeon Go, Semyung University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SMCOH-IM01
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: Temperature Change
Keywords: Temperature Change; Moxibustion; Warming effect
MeSH Terms: interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shingigu (Active Comparator): Treat with Shingigu
  Interventions: Device: Moxibustion
- Charcoal (Active Comparator): Treat with Charcoal
  Interventions: Device: Moxibustion

INTERVENTIONS:
Device: Moxibustion — Comparison of different kinds of moxibustion

SUMMARY:
The purpose of this study is to evaluate efficacy of Shingigu and Charcoal moxibustion scientifically and objectively.

DETAILED DESCRIPTION:
Moxibustion is traditional treatment that regulate circulation of Qi-blood by making the body warm to prevent and treat disease. Recently many kinds of moxibustion and moxibustion apparatus were developed. However evaluating efficacy of moxibustion is insufficient. Thus, there is need for objective evaluating about efficacy of moxibustion.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old

Exclusion Criteria:

* Hyperthyroidism
* Heart disease(Heart failure, angina pectoris, myocardial infarction)
* Uncontrolled hypertension (SBP>145mmHg or DBP>95mmHg)
* Severe renal disorder
* Severe liver disorder
* Diabetes Mellitus
* Female are in the duration of pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Temperature Change after moxa treatment | 30 minutes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hoyeon Go, O.M.D., Principal Investigator — Semyung University Chungju Hospital
Locations (1):
- Semyung University Chungju Hospital, Chungju, North Chungcheong, South Korea